CLINICAL TRIAL: NCT06854783
Title: A Phase 1, Open-Label, Multiple Dose Study to Assess the Pharmacokinetics, Safety, Tolerability, and Food Effect of MRX1 in Healthy Adults
Brief Title: Safety and Pharmacokinetics of Cannabidiol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tiamat Australia Pty Ltd (Industry)
Collaborators: Ananda Pharma plc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: MRX1-1-001
Record Dates: First submitted 2025-02-14; First posted 2025-03-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-07

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Low Dose (Experimental): Group A:
  Period 1 (Fasted): Cannabidiol at 2.5 mg/kg of body weight, administered twice daily (BID) for 5 days, with a single dose administered on the morning of Day 6 (n=10). All doses will be administered in a fasted state.
  Following a 14-day washout period, all participants will enter Period 2.
  Period 2 (Fed): Cannabidiol at 2.5 mg/kg of body weight, administered once on the morning of Day 21 following consumption of a standardised high fat, high calorie meal (n=10).
  Interventions: Drug: Cannabidiol
- Group B High Dose (Experimental): Group B
  Period 1 (Fasted): Cannabidiol at 7.5 mg/kg of body weight, administered BID for 5 days, with a single dose administered on the morning of Day 6 (n=10). All doses will be administered in a fasted state.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, safety, tolerability and food effect of investigational drug MRX1 in healthy adults.

DETAILED DESCRIPTION:
MRX1 is an oral solution containing cannabidiol.

The primary objective of this study is the assess the pharmacokinetic profile of MRX1 at two doses when administered twice daily in healthy adults. The secondary objectives are to assess the safety and tolerability of MRX1 and to characterise the effect of a high fat, high calorie meal on the pharmacokinetics of a single dose of MRX1.

A total of 20 healthy volunteers (10 male and 10 female) will be sequentially enrolled into 2 treatment groups, with 5 males and 5 females in each group.

The duration of the study is up to 52 days per participant for Group A and 37 days per participant for Group B, including screening and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide voluntary, written informed consent
* Males and females, aged 18 to 55 years inclusive at time of informed consent.
* Total body weight ≥50 kg and body mass index (BMI) between 18 and 32 kg/m2 inclusive.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening and Day -1.
* WOCBP must agree to the use a highly effective birth control (refer to Appendix 11.1) from Screening through 30 days following the last dose of study drug.
* Male participants must agree to use highly effective birth control including condom (refer to Appendix 11.1) from Screening through 90 days following the last dose of study drug. Male participants with female partners that are surgically sterile or post menopausal (defined as being amenorrhoeic for at least 12 months without an alternative medical cause), or male participants who have undergone sterilisation and have had testing to confirm the success of the sterilisation, may also be included and will not be required to use above-described methods of contraception. Male participants must also agree not to donate sperm up to 90 days following the last dose of study drug.
* Considered healthy, as determined by medical evaluation by the Investigator including medical history and physical examination.
* Vital signs after 5 minutes resting in supine position within the following ranges: Systolic blood pressure: 90 to 140 mmHg inclusive; Diastolic blood pressure: 40 to 90 mmHg inclusive; Heart rate: 40 to 100 bpm inclusive.
* Standard 12-lead ECG with parameters (average of triplicate readings) after 10 minutes in supine position within the following ranges: QRS <120 msec; QT <500 msec; QTc ≤450 msec (both genders); PR interval ≥120 to ≤220 msec.
* Negative tests for HBsAg, HBcAb (if HBsAg positive), anti-HCV, and HIV antibody at Screening (positive anti-HCV antibody allowed if HCV PCR is negative).
* Screening and Day -1 safety laboratory test values within normal ranges. Out of normal range values may be accepted by the Investigator if not considered clinically significant, with the exception of the following: ALT or AST >1.5 x upper limit of normal (ULN); Total, indirect, or direct bilirubin >1.5 x ULN. Participants with Gilbert's syndrome with indirect bilirubin outside of the normal range will be excluded from the study.
* Willing to refrain from consumption of alcohol as follows: Group A: for at least 48 hours prior to Screening, Day -1, and Day 20, and throughout the in-patient confinement periods and post-dose follow-up visits (consumption of alcohol is permitted during the outpatient washout period); Group B: for at least 48 hours prior to Screening and Day -1, and throughout the study.
* Willing to defer blood donations to a blood service for minimum of 30 days following the last dose of study drug.
* In the opinion of the Investigator, is willing and able to comply with and understand study requirements and be available for the required study visits.

Exclusion Criteria:

* Female participant who is pregnant or breastfeeding, or planning to become pregnant or breastfeed, or planning to donate ova during study participation.
* History or presence of a medical condition that, in the opinion of the Investigator, would interfere with the evaluation of the study drug or lead to increased risk of harm.
* Presence of any chronic medical condition requiring ongoing treatment.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks prior to Screening, as per Investigator judgement.
* Documented evidence of current or past cardiovascular disease including cardiac arrhythmias or family history of congenital long QT syndrome, Brugada syndrome, or unexplained sudden cardiac death.
* Any gastrointestinal surgery or condition or disease that could affect drug absorption, distribution, or excretion (e.g., gastrectomy, cholecystectomy, diarrhea, recurrent nausea/vomiting).
* History of malignancy of any organ system (other than localised basal cell carcinoma of the skin or in situ cervical cancer considered treated and cured), treated or untreated, within 5 years before Screening, regardless of if there is no evidence of local recurrence or metastases.
* History of schizophrenia, bipolar disorder psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis including generalised anxiety and obsessive-compulsive disorders. Hospitalisation within 5 years before Screening due to psychiatric illness or due to danger to self or others.
* Current use (or within the 3 months prior to Screening) of other cannabinoid or cannabis products.
* History of allergy or other adverse reaction to cannabinoid or cannabis products at any time in the past or known or suspected hypersensitivity to any of the components of the formulation.
* Current or recent (within 2 months prior to Screening) use of any tobacco or nicotine products (including e-cigarettes, vaping, or dipping) at >5 cigarettes per week or equivalent. Causal/social smokers (≤5 cigarettes per week or equivalent) are permitted.
* History of substance abuse disorder(s), as determined by the Investigator, within 5 years of Screening, including but not limited to alcohol, illicit drugs, and inappropriate use of prescription drugs.
* Positive urine drug test or alcohol breath test at Screening or Day 1, unless there is an explanation deemed acceptable by the Investigator and/or the participant tests negative upon re-test (one re-test permitted per scheduled time point).
* Use of any prescription medicines or marijuana within 14 days of Day -1 or use of any nonprescription medicines, supplements, or vaccines within 7 days of Day 1. Occasional (PRN) paracetamol (up to 2 g/day) or ibuprofen (up to 1.2 g/day) use may be permitted, at Investigator discretion. Hormonal contraceptives are permitted.
* Consumption of food and/or beverages containing Seville oranges or Seville orange juice, or grapefruit or grapefruit juice, or poppy seeds within 7 days prior to Day -1.
* Consumption of caffeine/xanthine products within 24 hours prior to Day -1.
* Use of any investigational drug within 30 days or <5 half-lives, whichever is longer, prior to first dose of study drug.
* Donation or receipt of any blood or blood products at a blood bank or donation centre within 30 days prior to Screening.
* Identified as a site employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members (i.e., immediate, husband, wife or de facto and their children, adopted or natural) of the site employees or the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration [Cmax] | Days 1, 6 and 21
  Maximum observed concentration for CBD, 7-OH-CBD and 7-COOH-CBD.
Pre-dose concentration [Ctrough] | From Day 2 to Day 6.
  Pre-dose concentration inclusive of CBD, 7-OH-CBD and 7-COOH-CBD.
Time to maximum observed concentration [Tmax] | Days 1 and 6.
  Time to maximum observed concentration of CBD, 7-OH-CBD and 7-COOH-CBD.
Area under the plasma concentration time curve 0-12 hours [AUC0-12] | Days 1, 6 and 21
  The area under the plasma concentration-time curve, from time 0 (time of dosing) to 12 hours for CBD, 7-OH-CBD and 7-COOH-CBD.
Area under the plasma concentration-time curve 0-24 [AUC0-24] | Day 1
  The area under the plasma concentration-time curve, from time 0 (time of dosing) to 24 hours for Group B and Group A, Period 1 for CBD, 7-OH-CBD and 7-COOH-CBD.

SECONDARY OUTCOMES:
Frequency and severity of adverse events | From Day 1 to end of study at Day 24.
  The frequency and severity of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI) as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No